CLINICAL TRIAL: NCT04519983
Title: Efficacy of SRT as Salvage Therapy in Patients With Brain Oligo-progression of EGFR-mutant Non-small Cell Lung Cancer After Failure of the Third-generation EGFR-TKIs: A Multicenter, Open Label, Phase II Clinical Study
Brief Title: Efficacy of SRT as Salvage Therapy in Patients With Brain Oligo-progression of EGFR-mutant Non-small Cell Lung Cancer After Failure of the Third-generation EGFR-TKIs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-BMSA
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer Stage IV
MeSH Terms: conditions — Lung Neoplasms | interventions — aumolertinib; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upfront TKI + Salvage SRT (Experimental): Patients With Brain metastases of EGFR-mutant Non-small Cell Lung Cancer should receive Aumolertinib as upfront treatment. SRT(32Gy/4fx) is given to progressive or recurrent intracranial lesions as salvage therapy after intracranial failure.
  Interventions: Drug: Aumolertinib Oral Tablet

INTERVENTIONS:
Drug: Aumolertinib Oral Tablet — Aumolertinib 110 mg p.o. qd+ SRT(32Gy/4fx)
  Other Names: Stereotactic Radiation Therapy

SUMMARY:
About 20%-40% of NSCLC patients develop intracranial metastases, and most clinical studies suggest that the survival of lung cancer patients will be significantly shortened once they develop intracranial metastases. EGFR tyrosine kinase inhibitors (EGFR-TKIs) remain the standard first-line therapy for patients with advanced EGFR-mutated NSCLC, including brain metastases(EGFR BMs). The survival rate of NSCLC patients with EGFR BMs was significantly improved compared with that of mutation-free patients. Third-generation EGFR-TKIs have unique advantages in the treatment of NSCLC BMs due to their improved blood-brain barrier permeability, and with the development of radiotherapy technology, stereotactic radiation therapy (SRT) has also demonstrated its remarkable qualities of high efficiency and low toxicity in a limited number of intracranial metastases. The clinical mechanisms of resistance to third-generation EGFR-TKIs are far more complex than those of first-generation TKIs, and the treatment paradigm for disease progression including intracranial progression is challenging. It would be interesting to design prospective clinical studies of patients with EGFR BMs treated with the third-generation TKIs followed by salvage SRT for oligo-progression. Therefore, the investigator designed this prospective, phase II clinical study of intracranial oligo-progression applied with stereotactic radiotherapy as salvage therapy in EGFR BMs patients after failure of the third-generation EGFR-TKIs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75.
2. Life expectancy exceeding 3 months.
3. Histologic or cytologic pathology confirmed non-small cell lung cancer. However, sputum cytology results alone are not acceptable. The cytology results of tracheal swabbing, tracheal irrigation fluid and needle aspiration are acceptable.
4. Investigators have confirmed the presence of at least one intracranial measurable lesion according to RECIST 1.1 criteria.
5. Patients with stage IV NSCLC with intracranial metastases at MR baseline.
6. Eastern Oncology Collaborative Group (ECOG) fitness status score of 0 or 1.
7. Genetic testing suggests EGFR driver gene positivity, which can be accompanied by other driver gene positivity.
8. Oligo-progression of intracranial tumors at the most recent evaluation following treatment with third- generation TKIs.
9. Good hematopoiesis, defined as an absolute neutrophil count ≥1.5 × 109/L, platelet count ≥100 ×109/L, blood erythropoietin ≥ 90 g/L [7 days without transfusion or erythropoietin (EPO-dependent).
10. Good liver function, defined as total bilirubin levels ≤ 1.5 times the upper limit of normal (ULN); inpatients without hepatic metastases, glutinous rice straw is used as a supplement.
11. Aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN; for patients with documented liver metastases. AST and ALT levels ≤5 times ULN.
12. Good renal function, defined as serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance ≥60 ml/min
13. (Cockcroft-Gault formula); less than 2+ urine protein on routine urinalysis, or 24-hour urine protein quantification <1 g.
14. Good coagulation, defined as an International Standardized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5times ULN; if the subject is receiving anticoagulant therapy, provided that the PT is within the intended range of use of the anticoagulant.
15. For female subjects of childbearing age, within 3 days prior to receiving the first study drug administration (Week 1, Day 1) A negative urine or serum pregnancy test is performed. If a negative urine pregnancy test cannot be confirmed, a blood pregnancy test may be ordered test.
16. High-performance contraception (i.e., methods with a failure rate of less than 1 per cent per year) for both male and female patients if there is a risk of conception.

Exclusion Criteria:

1. NSCLC EGFR driver gene negativity.
2. Patients who cannot be examined by MR.
3. Pathological examination of a mixture of small cell lung cancer components.
4. Currently participating in an interventional clinical research treatment or have received another investigational drug within 4 weeks prior to the first administration of the drug.
5. Use of third-generation TKIs or major surgical procedures within 3 weeks prior to the first dose of the drug.
6. Received palliative intracranial radiotherapy prior to first administration.
7. Presence of clinically active diverticulitis, abdominal abscesses, gastrointestinal obstruction.
8. Have received a transplant of a solid organ or blood system.
9. Presence of clinically uncontrollable pleural effusion/abdominal fluid.
10. Known severe allergic reaction (≥ grade 3) to TKIs.
11. Have not sufficiently recovered from toxicity and/or complications from any of the interventions prior to initiating treatment (i.e. ≤ grade 1 or at baseline, not including weakness or hair loss).
12. Diagnosis of other malignancies within 5 years prior to the first dose, with exceptions including radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radically resected carcinoma in situ.
13. Active infections that require systemic treatment.
14. The known existence of a mental illness or substance abuse condition that may affect compliance with the test requirements.
15. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive).
16. Evidence of a medical history or illness that could interfere with the results of the trial, prevent the subject from participating throughout the study, abnormal values for treatment or laboratory tests, or other circumstances that, in the opinion of the investigator, make enrollment unsuitable.
17. Breastfeeding women.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Intracranial objective response rate (iORR) | 2 years
  the rate at which intracranial lesions experience complete and partial remission compared to baseline
Intracranial progression-free survival (iPFS) | 2 years
  the time between receiving treatment, observing intracranial disease progression or occurrence of death from any cause, two orders of iPFS will be available in this study analysis. Patients who are still alive at the time of analysis will have the date of their last contact as the cut-off date.

SECONDARY OUTCOMES:
Overall survival (OS) | 2years
  the time between receiving treatment, observing disease progression at any site, or occurrence of death from any cause, there will be two orders of PFS available for analysis in this study. Patients who are still alive at the time of analysis will have the date of their last contact as their cut-off date.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China